CLINICAL TRIAL: NCT06212531
Title: The Papuan Indigenous Model of Voluntary Clinical Male Circumcision
Brief Title: Papuan Indigenous Model of Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Atma Jaya Catholic University of Indonesia (Other)
Responsible Party: Principal Investigator, Robert Bailey, Distinguished Professor Emeritus, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0661; R21AI155926 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: HIV Infections
Keywords: HIV Prevention; Male circumcision; Papua Indonesia
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Observational study of recruitment of young Papuan men who volunteer for medical male circumcision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Medical male circumcision using standard surgical technique. — Medical male circumcision using the WHO standard technique followed by examination of wound healing and behavioral risk assessment.

SUMMARY:
The purpose of the study is: AIM 1: To engage Papuan community members to explore acceptability, barriers and facilitators for introducing a school-based age and culturally appropriate, comprehensive VMMC intervention to reduce HIV incidence in the Papuan population. AIM 2: To assess the capacity of the community health system to meet international criteria for safe comprehensive VMMC services and to ensure the availability of resources and training necessary to meet these criteria in selected clinics. AIM 3: To design the PIM of school-based adolescent VMMC based on information collected in Aims 1 and 2 and in consultation with a community advisory board, the Ministry of Health and the Ministry of Education. AIM 4: To pilot-test the school-based PIM Intervention of VMMC with 400 boys ages 12-18 years at two HIV high-risk Papuan locations: the Nabire and Jayapura. Primary outcomes are the proportion of adolescent males exposed to school-based PIM VMMC educational and informational sessions who get circumcised and surgical event safety. Secondary outcomes are satisfaction by adolescent males and parents, any sexual activity within 6 weeks after circumcision, changes in sexual risk behaviors between base-line and 12 weeks after circumcision, and perceptions of providers regarding MC training and implementation, ease of device use, and challenges encountered.

ELIGIBILITY:
Inclusion Criteria:

* Resident of either Nabiri or Jayapura Districts of Papua, Indonesia. Able to provide informed consent if over 17 and parental consent and personal assent if less than 18.

Focus group and interview participants had to be either a parent, boy or girl between 12-18, teacher or administrator, or community leader.

To be eligible for circumcision, a boy had to be uncircumcised, age 15 years or above, and not show signs or symptoms of an STI or any penile abnormality (e.g., hypospadias, phimosis) that made him clinically ineligible for circumcision.

Exclusion Criteria:

* Unable to provide informed consent or assent. Any medical condition indicating should not undergo circumcision.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of male exposed to intervention who get circumcised. | 6 months
  The proportion of males who are recorded attending school-based PIM VMMC educational and informational sessions who are recorded as getting circumcised and at community health clinics.

SECONDARY OUTCOMES:
Levels Satisfaction | 4 months
  Levels of satisfaction by adolescent males and parents measured through face-to-face interview questionnaires using a five item likert scale.
Sexual Behavior | 4 months
  Sexual activity within the first 6 weeks after circumcision measured by face-to-face interview, including whether or not they have had sex, number of sex partners and condom use.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, School of Public Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No